CLINICAL TRIAL: NCT05566301
Title: MULTIcentric Study About RESistance to CLOpidogrel in Dual Antiplatelet Therapy for Carotid Stenting
Brief Title: Multicentric Study on Clopidogrel Resistance in DAPT for CAS (MULTI-RESCLOSA)
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Daniela Mazzaccaro, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: MULTI-RESCLOSA v.1 16-2-21
Record Dates: First submitted 2022-09-28; First posted 2022-10-04 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Clopidogrel, Poor Metabolism of; Carotid Stenosis
Keywords: clopidogrel resistance; carotid artery stenting; carotid stenosis; dual antiplatelet therapy; ticagrelor
MeSH Terms: conditions — Carotid Stenosis | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clopidogrel: Patients who undergo carotid stenting and dual antiplatelet therapy with ASA + clopidogrel and whose aggregometry test shows correct response to the effect of clopidogrel
  Interventions: Drug: Clopidogrel
- Ticagrelor: Patients who undergo carotid stenting and dual antiplatelet therapy with ASA + clopidogrel and whose aggregometry test shows incorrect response to the effect of clopidogrel, therefore therapy is switched to ASA + ticagrelor
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — All patients will undergo carotid stenting and dual antiplatelet therapy with ASA + clopidogrel
  Groups: Clopidogrel
Drug: Ticagrelor — All patients will undergo carotid stenting and dual antiplatelet therapy with ASA + clopidogrel
  Groups: Ticagrelor

SUMMARY:
Spontaneous prospective observational multicentre pharmacological study that aims to evaluate whether, from a statistical point of view, there is a significant difference between the use of Ticagrelor in "non-responders" patients to Clopidogrel undergoing carotid stenting and Clopidogrel in "responders" undergoing carotid stenting, in the onset of death and major adverse cardiovascular events (MACE) and bleeding events, 1 and 3 months after the procedure. Furthermore, the study aims to evaluate the possible preoperative clinical and pharmacological factors most associated with the phenomenon of resistance to Clopidogrel.

Inclusion criteria:

The data will be collected on adult patients (age> 18 years) who have given their consent to participate in the study, belonging to the U.O. of Vascular Surgery of the IRCCS Policlinico San Donato and the U.O. of Vascular Surgery of the participating centers and there subjected to the treatment of carotid stenosis by stenting technique.

Exclusion criteria:

Those patients who are minors, who have not given their consent to participate in the study, or who have carotid stenosis not susceptible to intervention by stenting will be excluded from the study. Pregnant or lactating women will also be excluded from the study (such as situations in which carotid stenting is contraindicated regardless of the execution of the study).

DETAILED DESCRIPTION:
Patients' records will be reviewed for clinical data (age, sex, height and weight), the presence of cardiovascular risk factors (diabetes mellitus, hypertension, dyslipidemia, smoking habits, coronary artery disease, chronic obstructive pulmonary disease), features of the carotid plaque (type of plaque and degree of carotid stenosis, according to ECST measurement), and status of the contralateral carotid artery. The occurrence of preoperative neurologic symptoms within the previous 6 months will also be recorded, as evaluated by the neurologist.

Preoperative and postoperative drug intake will be investigated, with particular attention to statins, beta blockers, angiotensin-converting enzyme (ACE) inhibitors, antiplatelet therapy and anticoagulant therapy.

Laboratory data such as serum creatinine, platelet counts, Red blood cell Distribution Width (RDW), Prothrombin Time (PT), International Normalized Ratio (INR), activated Partial Thromboplastin Time (aPTT) and ratio will be also assessed.

After operation, patients will be followed up three times in the first year (at 1 month, 6 months, and 12 months) and annually thereafter, using ultrasound. An angio-Computed Tomography scan will be required when complications were detected at ultrasound examination. During follow-up, data will be collected about the occurrence of death, stent thrombosis, cerebrovascular events, cardiac events, major haemorrhagic events.

Determination of the effectiveness of antiplatelet drugs The effectiveness of antiplatelet drugs will be evaluated through the impedance aggregometry test, conducted with the Multiplate® platelet function analysis V2.03.11 (Roche, Basel, Switzerland).

Multiplate® technology is based on the principle of electrical impedance aggregometry for the determination of platelet function on whole blood.

The instrument has five independent channels for parallel measurement and is connected to a computer equipped with specific software for the analysis and display of results in real time.

The blood and reagents are placed in a disposable cuvette containing two pairs of electrodes, representing two independent sensor units for a duplicate measurement. The platelets activated by the specific agonist adhere to the metal surface of the sensors, forming an insulating layer and increasing the electrical impedance between the electrodes. The change in impedance due to adhesion and platelet aggregation is represented as a function of time. The area included within the aggregation curve, used to measure aggregation, is expressed in arbitrary aggregation units (U). Since the change in impedance is measured simultaneously on two sensors, the results of each test are expressed as the average value of the two aggregation curves obtained.

Blood sampling to assess platelet aggregation was performed at the patient's hospitalization (in the event that he was already taking clopidogrel), or at least 6 hours after the start of antiplatelet therapy with clopidogrel.

The aggregometry test evaluates the efficacy of salicylates (ASPI-test, aggregation with the use of arachidonic acid: normal reference values 71-115 U) and the efficacy of drugs that act on the adenosine diphosphate (ADP) receptor such as thienopyridines. (ADP-test, ADP-triggered aggregation: normal reference values 57-113 U), compared to the positive control for platelet reactivity by the thrombin-receptor activating peptide (TRAP)-6 (TRAP-test: normal reference values 84-128 U).

In particular, 4 mL of either arterial or venous whole blood will be collected in a tube containing the specific anticoagulant hirudin. Three hundred µL of whole blood diluted with 300 µL of physiological solution will be placed in a disposable cuvette with the aid of an automatic pipette, and left to incubate at 37 ºC for 3 minutes. After incubation, a specific agonist will be added for the required exam. The platelet aggregation value will be measured over the next 6 minutes.

The effectiveness of clopidogrel is defined by the evidence of ADP-test which results to be under normal reference values, otherwise the patient is considered to be resistant to the effect of the drug.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age> 18 years)
* patients who have given their consent to participate in the study, belonging to the U.O. of Vascular Surgery of the IRCCS Policlinico San Donato and the U.O. of Vascular Surgery of the participating centers and subjected to the treatment of carotid stenosis by stenting technique.

Exclusion Criteria:

* underage patients
* patients who have not given their consent to participate in the study,
* patients who have carotid stenosis not susceptible to intervention by stenting
* pregnant or lactating women (such as situations in which carotid stenting is contraindicated regardless of the execution of the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo carotid stenting for a significant carotid stenosis and who are treated with dual antiplatelet therapy using ASA + clopidogrel
Sampling Method: Non-Probability Sample
Enrollment: 1140 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | 1 month
  Outpatient visit
Death | 3 months
  Outpatient visit
MACE | 1 month
  Major Adverse Cardiovascular Events, Outpatient visit
MACE | 3 months
  Major Adverse Cardiovascular Events, Outpatient visit
Occurrence of major hemorrhagic events | 1 month
  Outpatient visit
Occurrence of major hemorrhagic events | 3 months
  Outpatient visit

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huibers A, Halliday A, Bulbulia R, Coppi G, de Borst GJ; ACST-2 Collaborative Group. Antiplatelet Therapy in Carotid Artery Stenting and Carotid Endarterectomy in the Asymptomatic Carotid Surgery Trial-2. Eur J Vasc Endovasc Surg. 2016 Mar;51(3):336-42. doi: 10.1016/j.ejvs.2015.11.002. Epub 2015 Dec 21. PMID 26717867
- [Background] Ricotta JJ, Aburahma A, Ascher E, Eskandari M, Faries P, Lal BK; Society for Vascular Surgery. Updated Society for Vascular Surgery guidelines for management of extracranial carotid disease. J Vasc Surg. 2011 Sep;54(3):e1-31. doi: 10.1016/j.jvs.2011.07.031. PMID 21889701
- [Background] Bertrand ME, Rupprecht HJ, Urban P, Gershlick AH; CLASSICS Investigators. Double-blind study of the safety of clopidogrel with and without a loading dose in combination with aspirin compared with ticlopidine in combination with aspirin after coronary stenting : the clopidogrel aspirin stent international cooperative study (CLASSICS). Circulation. 2000 Aug 8;102(6):624-9. doi: 10.1161/01.cir.102.6.624. PMID 10931801
- [Background] Hurst NL, Nooney VB, Raman B, Chirkov YY, De Caterina R, Horowitz JD. Clopidogrel "resistance": pre- vs post-receptor determinants. Vascul Pharmacol. 2013 Nov-Dec;59(5-6):152-61. doi: 10.1016/j.vph.2013.10.002. Epub 2013 Oct 16. PMID 24140755
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Park MW, Kim CJ, Kim MC, Choo EH, Hwang BH, Park CS, Kim HY, Yoo KD, Jeon DS, Jeong MH, Seung KB, Ahn Y, Chang K. A prospective, multicentre, randomised, open-label trial to compare the efficacy and safety of clopidogrel versus ticagrelor in stabilised patients with acute myocardial infarction after percutaneous coronary intervention: rationale and design of the TALOS-AMI trial. EuroIntervention. 2021 Feb 19;16(14):1170-1176. doi: 10.4244/EIJ-D-20-00187. PMID 32718912